CLINICAL TRIAL: NCT06077084
Title: High Versus Moderate Intensity Neck Strengthening Treatment for Improving Disability, Neck Muscle Morphometry and Composition in Non-Specific Chronic High Versus Moderate Intensity Neck Strengthening Treatment for Improving Disability, Neck Muscle Morphometry and Composition in Non-Specific Chronic Neck Pain
Brief Title: Neck Strengthening in Non-Specific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universite de La Reunion (Other)
Collaborators: Le Mans Universite (Other)
Responsible Party: Principal Investigator, Francis Grondin, PhD-student, physiotherapist, Universite de La Reunion
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CERVIR
Record Dates: First submitted 2023-06-06; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate intensity (Active Comparator)
  Interventions: Other: Physiotherapy
- High intensity (Active Comparator)
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — 4months with multimodal physiotherapy. 2 sessions/week. Sessions consisted of two sessions of 1 hour per week, focusing on neck and arm movements. Each session included education and manual therapy (20 minutes), and exercises targeting neck extensors, flexors, and shoulder girdle muscles (40 minutes).
  Low-intensity neck resistance training :
  Participants have to perform arm, neck flexors and extensors exercise. motor control exercises focusing on deep neck muscles, slow dynamic and static contractions (10 to 20 seconds) with low resistance using TheraBand and weights ranging from 0.5 kg to 1 kg.
  High-Intensity Neck resistance training :
  neck flexors exercise, neck extensors exercise, and one exercise for shoulder/upper limb. static contractions (10-seconds) and dynamic neck movements using a handheld biofeedback dynamometer or weights from 50% to 80% of the 1-repetition maximum

SUMMARY:
This study aims to investigate the effects of exercise interventions on neck muscle morphometry and composition in individuals with chronic non specific neck pain. The participants will be randomly assigned to either a moderate intensity or a high intensity neck strengthening program. The primary outcomes include neck disability. Secondary outcomes include changes in muscle volume and fat infiltration in the neck muscles measured using MRI, pain intensity, anxiety, and depression. The results of this study will contribute the future rehabilitation strategies.

DETAILED DESCRIPTION:
Chronic neck pain is a prevalent condition that significantly affects the quality of life for many individuals. It has been observed that individuals with chronic neck pain may experience alterations in muscle composition, including changes in muscle volume and the presence of fat infiltration. Exercise interventions have shown promise in improving muscle function and reducing pain in this population.

Objective:

The objective of this randomized controlled trial is to investigate the effects of two different exercise interventions on the disability and muscle composition in individuals with chronic non specific neck pain. The study aims to compare the outcomes of a moderate intensity neck strengthening program and a high intensity neck strengthening program.

Methods:

Participants will be recruited and randomly assigned to either the moderate intensity neck strengthening (MINS) group or the high intensity neck strengthening (HINS) group. The exercise interventions will be supervised by qualified physiotherapists and will consist of targeted exercises specifically designed to strengthen the neck muscles.

Outcomes :

Magnetic resonance imaging (MRI), Neck Disability Index (NDI), pain intensity, psychological measures such as anxiety and depression using validated questionnaires.

Data analysis :

Pre- and post-intervention measurements within each group and examining the between-group differences.

Conclusion:

This study aims to provide valuable insights into the effects of different exercise interventions on the disability an neck muscle morphometry/composition in individuals with chronic non specific neck pain. The study aims to enhance the understanding of the underlying mechanisms and potential benefits in this population. The findings may contribute to the development of targeted rehabilitation strategies that can effectively improve muscle function and reduce pain in individuals with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* have experienced chronic non-specific neck pain for at least three months, exhibit symptoms triggered by neck movement, and score at least 20% on the Neck Disability Index questionnaire

Exclusion Criteria:

* history of head or neck surgery or fracture, rheumatoid or metabolic disease, inability to understand or write in French, significant trauma such as a car accident, previous or current neoplasm, known psychiatric conditions like bipolar disorder, current pregnancy for women, clinical or radiological neurological features, cardiovascular or respiratory conditions, and drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Neck disability Index score | At inclusion and 2 weeks after the 4-months treatment
  questionnaire, a higher score means worst disability

SECONDARY OUTCOMES:
Neck muscle volume of multifidus, spinalis cervicis longus colli, levator scapulae, spinalis capitis, splenius capitis, sternocleidomastoideus, | At inclusion and 2 weeks after the 4-months treatment
  Muscle volume measured with magnetic resonance imagery, a higher volume could means better improvement
Fat infiltration in neck muscle morphometry of multifidus, spinalis cervicis longus colli, levator scapulae, spinalis capitis, splenius capitis, sternocleidomastoideus. | At inclusion and 2 weeks after the 4-months treatment
  % of fat infiltration measured by magnetic resonance imagery, a higher score means worst fat infiltration
Pain | At inclusion and 2 weeks after the 4-months treatment
  Numeric Pain Rating Scale of neck pain, a better score means worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Université de la Réunion, Le Tampon, La Réunion, Reunion

IPD SHARING:
Plan to Share IPD: No
Study Protocol & Informed Consent Form will be shared